CLINICAL TRIAL: NCT02453295
Title: Testing an Intervention to Foster Hope for Cancer Survivors With Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ottawa (Other)
Collaborators: University of New Brunswick (Other); McGill University (Other); Horizon Health Network (Other); New Brunswick Health Research Foundation (Other)
Responsible Party: Principal Investigator, Roanne Thomas, Canada Research Chair/Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: HopePilot
Record Dates: First submitted 2015-05-19; First posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Mastectomy Related Lymphedema; Lymphedema of Upper Limb; Lymphedema of Lower Extremity
Keywords: Lymphedema; Arm Disability; Cancer Survivorship; Intervention
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): The IG will meet weekly for 2 hours for 8 weeks. All workshops will be recorded and transcribed, then analyzed qualitatively. Administration of questionnaires (Meaning of Illness, MIQ; Herth Hope Index, HHI; Short Form 12, SF-12; Lymphedema Quality of Life, LYMQOL) will take place over the phone. The questionnaires will be administered 3 days prior to workshop 1 (T0), between workshop 4 and 5 (T1), and 3 days following the completion of the intervention (T2). The questionnaires will also be administered at 4 weeks post-intervention (T3) and 8 weeks (T4) post-intervention. All participants will also complete a demographic questionnaire at T0, developed in S2.
  Interventions: Behavioral: Intervention Group
- Comparison Group (No Intervention): The CG will receive LE treatment as usual, without the hope intervention. They will be administered the same questionnaires (by phone) as the IG at the same timepoints. Potential participants (n=46) will be screened based MIQ. The individuals scoring in the top ~30% (n=16) will be excluded from the study. The remaining 30 individuals scoring the lowest level of hope will be admitted into the study.

INTERVENTIONS:
Behavioral: Intervention Group — The IG will meet weekly for 2 hours for 8 weeks. Administration of questionnaires (Meaning of Illness, MIQ; Herth Hope Index, HHI; Short Form 12, SF-12; Lymphedema Quality of Life, LYMQOL) will be completed by phone at all timepoints. The questionnaires will also be administered at 4 weeks post-intervention (T3) and 8 weeks (T4) post-intervention. All participants will also complete a demographic questionnaire at T0, developed in S2 as well as a Workshop Evaluation 2 days following the final workshop (T2).
  Arms: Intervention Group

SUMMARY:
The specific objectives and research questions of the proposed study are:

1. a. Administer a group rehabilitation intervention to address loss and foster hope in 30 participants with upper and lower limb SLC --15 in an intervention group (IG), 15 in a control group (CG) at each of two research sites (Montreal, QC and Saint John, NB) for a total sample size of 60. Data about its impact will be collected by means of audiorecording 8 intervention workshops at each site and administering questionnaires (multiple timepoints).

   b. Test the intervention - Main hypothesis: The intervention group will show improvements in psychosocial well-being.
2. Assess feasibility (e.g., review our accrual strategies, randomization of participants, and data collection) via the completion of process logs.

DETAILED DESCRIPTION:
This mixed methods pilot study builds on completed interviews with 13 participants in 2012 (Study 1, S1) and delivery of a community-based intervention to 13 participants in 2013 (over 2 days; Study 2, S2). The proposed research draws on these two studies, S1 (REB#H-05-12-04) and S2 (REB#H-05-12-04B), both of which were approved by the uOttawa REB. S2 included the same intervention as the one proposed herein, but in a compressed format. It was delivered in Ottawa, with positive feedback received from all 13 participants.

Administration of the intervention will draw upon the team members' expertise (Hamilton, Hack) with interventions for people with cancer, a program of research in hope interventions, and Thomas' work with women with breast cancer related LE as well as S1 and S2. The intervention will follow a group-based workshop format. The intervention workshops will be offered weekly over 8 sessions (2 hours per session, one per week). After an introductory workshop, the second session will involve viewing the video, created by PI Thomas interviewing men and women who have lymphedema and group discussion of its themes, based on the principles of video modelling (e.g., how do participants' experiences, hope strategies compare?). This is an approach used successfully in other areas of research with marginalized peoples.

Our program will follow Herth's theoretical foundations and goals (e.g., identifying support systems, developing plans to maintain hope in the future) along with established approaches to supportive care in chronic illnesses and LE international best practice guidelines. Briefly, workshops include modules addressing the building of a supportive community; orienting to hope and identifying threats to hope/coping; positive self-talk and affirmations; creative practices for exploring experiences and hope; and identifying and mobilizing resources. The modules also incorporate the completion and discussion of creative projects (e.g., writing exercises), mini-lectures by rehabilitation professionals, and SLC resources. All of these components were reviewed positively (satisfactory or above) by the majority of participants in S2. All activities are drawn from Herth's intervention, prior research, and the success of S2. This content was approved by the uOttawa REB, as noted previously. Four questionnaires administered to the IG/CG will be used to assess the potential impact of the intervention. Please see Study Protocol for summary of data collection.

SUMMARY OF QUESTIONNAIRES

1. The Meaning of Illness Questionnaire, (MIQ) Factor II and IV: Factor II addresses loss, stress, and function. Factor IV addresses hope as well as positive attitude and motivation. These 2 factors will be used to screen participants prior to the study.

   The full version of the MIQ will be administered at all timepoints once the study begins, along with the other questionnaires.
2. The Herth Hope Index (HHI) is a 12-item (4 point) Likert scale that delineates 3 factors of hope: a) temporality & future, b) positive readiness & expectancy, and c) interconnectedness. (32) Summative scores range from 12-48, with a higher score denoting greater hope. The HHI was piloted in and deemed to be acceptable in S2. Participants encountered few difficulties with completion.
3. Short Form 12, (SF-12): is a QOL scale that measures seven concepts, including physical functioning, role limitations due to health problems, and social functioning. It is a shorter but valid alternative to the SF 36 and includes psychological aspects of illness (e.g., feeling energetic) not addressed by other instruments but relevant to S1 and S2 participants ;
4. Lymphedema Quality of Life, LYMQOL: is a validated measure for the impact of UL/LL LE. (110) The instrument includes 28 UL items and 27 LL items for LE. Importantly, questions address physical LE symptoms, emotional impact, and activities of daily living.
5. Demographic and Symptoms Questionnaire - contains 16 questions pertaining to age, family size, income and employment, and SLC symptoms. This questionnaire will only be administered at T0.

DATA COLLECTION

The IG will meet weekly for 2 hours for 8 weeks. All workshops will be recorded and transcribed, then analyzed qualitatively. The questionnaires (Meaning of Illness, MIQ; Herth Hope Index, HHI; Short Form 12, SF-12; Lymphedema Quality of Life, LYMQOL) will be administered by phone at the following timepoints: approximately 3 days prior to the first workshop (T0), between workshop 4 and 5 (T1) and approximately 3 days following the final workshop (T2). The questionnaires will also be administered at 4 weeks post-intervention (T3) and 8 weeks (T4) post-intervention. All participants will also complete a demographic questionnaire at T0, developed in S2.

For the Montreal site, the intervention (and post intervention data collection) will be administered by Chad Hammond (PhD, Psychology), a postdoctoral fellow who has worked extensively with cancer survivors. For Saint John, a qualified postdoctoral fellow will be hired by Co-PI Hamilton through the University of New Brunswick. Both will be trained by the Co-PIs.

The CG will receive LE treatment as usual, without the hope intervention. Participants will be asked to refrain from joining similar, group-based workshops over the duration of the intervention. The measures will be administered the same questionnaires (by phone) as the IG at the same timepoints. Montreal and Saint John (ethics approval to be obtained from McGill U, UNB, and Health Horizon) has been selected for the current proposal as workshops were already completed in Ottawa (S2).

At each site (Montreal and Saint John) potential participants (n=46) will be screened for eligibility based on Factors II and IV from the MIQ. The individuals scoring in the top ~30% (n=16) in terms of hope will be excluded from the study. The remaining 30 individuals scoring the lowest level of hope as per the MIQ will be admitted into the study. This initial appraisal will be brief, conducted over the phone, and therefore not too burdensome for potential participants. The investigators have chosen not to administer the full version of the MIQ (or other instruments) in order to screen efficiently and avoid potential practice and carryover effects in the administration of our other outcome measures. Towers (Montreal Co-I) and Tilley (Saint John Co-I) will approach potential participants in their LE clinics and their names/contact information will be forwarded to Dr. Chad Hammond, postdoctoral fellow (PDF) at the University of Ottawa for screening and randomization to the IG or CG.

Questionnaires: S1 data and prior SLC research informs the selection of hope as the main outcome measure, using the HHI.

EVALUATING THE INTERVENTION

The impact of the intervention will be measured by assessing changes in outcomes over an 2-month period. Questionnaires will be administered at intake (T0), midpoint (i.e., between workshop 4 and 5, T1), 3 days post-completion of the 8-week program (T2), 4 weeks post-intervention (T3), and 8 weeks post-intervention (T4). All participants will also complete a demographic questionnaire (T0), developed in S2. IG data will be collected via phone at all timepoints. A workshop evaluation form will also be administered to the IG at T2.

CG data will be collected by phone at all timepoints (however, the workshop evaluation is irrelevant to the CG and will not be collected). The follow-up period is consistent with studies in systematic reviews and meta-analyses of psychosocial interventions for people with cancer. Participants who leave the study early will be asked to complete a telephone exit interview to explore and moderate completion (acceptability) issues for future programming and research. Notes from these interviews will be compiled as part of the assessment of feasibility.

ASSESSING FEASIBILITY

S2 used a convenience sample, with posters displayed in clinicians' offices. Based on this limited advertising and resulting timely accrual the investigators are confident that the investigators can achieve our target of 30 participants within 12 weeks as the investigators will be approaching SLC patients directly through 2 LE clinics (Montreal, QC and Saint John, NB). Using this screening measure, the investigators will endeavour to enroll equal numbers of men and women as well as those with UL/LL. The # approached, # meeting inclusion criteria, and reasons for declining will be documented. As this is a pilot, the investigators will proceed to the intervention phase whether or not the groups represent equal numbers of men/women and upper limb (UL)/lower limb (LL). However, data gathered will be used to inform adjustments that might be required for a future full trial. Consistent with RCTs and in preparation for a full trial, a participant flow diagram (# assessed for eligibility, # excluded, # refuse to participate, # randomized, # allocated to IG and CG, # lost to follow-up, # discontinued, # analyzed, # excluded from analysis) will summarize statistics for recruitment and retention. Participants will be considered to have left the intervention when they are absent from 25% (2/8) of the workshops and will be asked to complete a short exit interview by telephone.

To assess the feasibility (and acceptability) of data collection, the investigators will address adherence to timepoints and barriers and facilitators to data collection. At the conclusion of the pilot, the impact of the intervention will be examined with an assessment of timeline data to determine whether all timepoints are feasible. If more than 50% of the sample requires more than 3 points of contact (phone and/or email) to schedule data collection, our team will modify the study design for a subsequent proposal (e.g., increase # of potential participants). Adherence to timepoint data will be generated through completion of a process log documenting dates of data collection for each participant as well as the # of points of contact required to schedule data collection. Descriptive statistics (frequencies, means, SD) will be generated to assess the feasibility of the timelines. Based on the data generated, timelines will be reviewed and adjusted if necessary before our subsequent CIHR proposal. Survey completion rates will be calculated, and % missing data will be noted. To provide additional data about acceptability, as in S2, IG participants will be encouraged to write notes on the hard copies of surveys (3 days prior Workshop 1 - T0; Intervention midpoint/between Workshop 4 and 5 - T1; Intervention completion/3 days following Week 8 - T2) to indicate any issues. These data will be transcribed, compiled, and analyzed. All of the above data will be triangulated to assess data collection feasibility.

ELIGIBILITY:
Inclusion:

* men and women who are 18 years of age or older;
* who have been diagnosed with UL or LL SLC a minimum of 3 months prior to data collection;
* who are in the management phase of SLC treatment at the time of enrolment;
* are English speaking;
* are able to consent.

Exclusion:

* being in the active phase of LE treatment. Because this type of acute care involves intensive and time-consuming treatment, which would make participation in the proposed research extremely challenging, we will enroll only men and women who are in the management phase of treatment.
* non-English speaking. Non-English speaking participants will be excluded given time and resource constraints. In our recent qualitative study of SLC, no non-English speaking potential participants from Ottawa expressed an interest in the study. Future research (to expand the pilot intervention, if successful) will be bilingual.
* As noted previously individuals scoring in the top ~30% (n=16) in terms of hope according to the MIQ, will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Adjustment to illness as per the Meaning of Illness (MIQ) tracked at 5 timepoints over 16 weeks | T0 - beginning (3 days prior to 1st workshop); T1 - midpoint; T2 - endpoint (3 days following final workshop); T3 - 4 weeks post-intervention; T4 - 8 weeks post-intervention
  Factor II and IV: Factor II addresses loss, stress, and function. Factor IV addresses hope as well as positive attitude and motivation. These 2 factors will be used to screen participants prior to the study.
  The full version of the MIQ will be administered at all timepoints once the study begins, along with the other questionnaires.
Level of hope as per the Herth Hope Index (HHI) tracked at 5 timepoints over 16 weeks | T0 - beginning (3 days prior to 1st workshop); T1 - midpoint; T2 - endpoint (3 days following final workshop); T3 - 4 weeks post-intervention; T4 - 8 weeks post-intervention
  12-item (4 point) Likert scale that delineates 3 factors of hope: a) temporality & future, b) positive readiness & expectancy, and c) interconnectedness.32 Summative scores range from 12-48, with a higher score denoting greater hope. The HHI was piloted in and deemed to be acceptable in S2. Participants encountered few difficulties with completion.
Quality of life as per the Short Form 12, (SF-12) tracked at 5 timepoints over 16 weeks | T0 - beginning (3 days prior to 1st workshop); T1 - midpoint; T2 - endpoint (3 days following final workshop); T3 - 4 weeks post-intervention; T4 - 8 weeks post-intervention
  Quality of Life (QOL) scale that measures seven concepts, including physical functioning, role limitations due to health problems, and social functioning. It is a shorter but valid alternative to the SF 36 and includes psychological aspects of illness (e.g., feeling energetic) not addressed by other instruments but relevant to S1 and S2 participants
Impact of lymphedema as per the Lymphedema Quality of Life (LYMQOL) tracked at 5 timepoints over 16 weeks | T0 - beginning (3 days prior to 1st workshop); T1 - midpoint; T2 - endpoint (3 days following final workshop); T3 - 4 weeks post-intervention; T4 - 8 weeks post-intervention
  Validated measure for the impact of UL/LL LE. The instrument includes 28 UL items and 27 LL items for LE. Importantly, questions address physical LE symptoms, emotional impact, and activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Hammond, PhD, Study Director — University of Ottawa